CLINICAL TRIAL: NCT01714882
Title: Stress Management for Couples With Infertility Undergoing In Vitro Fertilization (IVF)
Brief Title: Stress Management for Couples Undergoing In Vitro Fertilization (IVF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amit Sood (Other)
Responsible Party: Sponsor-Investigator, Amit Sood, Associate Professor of Medicine, Consultant - General Internal Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-007272
Record Dates: First submitted 2012-10-18; First posted 2012-10-26 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Infertility
Keywords: Infertility; In Vitro Fertilization (IVF); Stress Management; Stress Reduction
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress Management & Resiliency Training (Experimental): The couples in this group will attend the SMART in-person training class at the beginning of the study and will be taught a structured relaxation program.
  Interventions: Behavioral: Stress Management & Resiliency Training
- Stress Management DVD (Active Comparator): The couples in this group will receive a Mayo Clinic Stress Management DVD.
  Interventions: Behavioral: Stress Management DVD

INTERVENTIONS:
Behavioral: Stress Management & Resiliency Training — The couples in this group will attend the SMART in-person training class at the beginning of the study and will be taught a structured relaxation program.
  Arms: Stress Management & Resiliency Training
Behavioral: Stress Management DVD — The couples in this group will receive a Mayo Clinic Stress Management DVD.
  Arms: Stress Management DVD

SUMMARY:
The investigators are trying to determine stress management strategies in couples undergoing In Vitro Fertilization (IVF).

DETAILED DESCRIPTION:
The investigators are trying to determine two different stress management techniques in couples undergoing IVF. One arm will be randomized to learning these techniques by themselves by watching and following instructions on a digital video disc (DVD). The other arm will have an in-person class that will teach the couples different stress reduction techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women with clinical infertility, either primary or secondary, who are recommended for IVF for the first time as part of their treatment for infertility
* Women with a partner, and both are willing to provide consent for study participation as a couple
* Couples that can be reached by telephone for follow-up

Exclusion Criteria:

* Women less than 18 years of age
* Women equal or greater than 40 years of age
* Women with a history of recurrent pregnancy loss
* History of current or recent psychotic episode within past 6 months for either the woman or her partner
* Couples needing a interpreter for their clinical encounter

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change of Scores from questionnaires from baseline to 6 and then 12 weeks | Baseline, 6 and 12 weeks after randomization
  Primary outcome measure will be comparison of pre- and post-stress reduction treatment questionnaire scale scores.

SECONDARY OUTCOMES:
Clinical Pregnancy rate | 12 months after randomization
  Clinical pregnancy rate: which is defined as seeing a gestational sac in the uterus with a fetal pole that has a heart beat.

OTHER OUTCOMES:
Clinical or biochemical miscarriage | 12 months after randomization
  Miscarriage will be defined as a biochemical or clinical miscarriage. A biochemical miscarriage will include a rise and then subsequent fall in beta human chorionic gonadotrophin (BhCG) to less than 5 IU/L. A clinical miscarriage will be defined as vaginal bleeding with passage of products of conception recognized as products of conception by histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, MD, Principal Investigator — Mayo Clinic; Zaraq Khan, MBBS, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States